CLINICAL TRIAL: NCT00104533
Title: Effectiveness of Magnetic Therapy on Pain Intensity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Javeriana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1753; 1203-04-16295
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2005-03

CONDITIONS: Postoperative Pain
Keywords: Static magnetic therapy; Pain; Analgesia; Opioids
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

INTERVENTIONS:
Device: Magnets

SUMMARY:
Static magnetic therapy is increasingly used to alleviate pain; however, its efficacy has not been determined yet.

The aims of this proposal are to evaluate the effect of magnetic therapy on pain intensity levels, opioid requirements, and opioid side effects.

DETAILED DESCRIPTION:
Static magnetic therapy is increasingly used to alleviate pain; however, its efficacy has not been determined yet. The aims of this proposal are to evaluate the effect of magnetic therapy on pain intensity levels, opioid requirements, and opioid side effects.

A randomized, double blind, controlled trial is proposed. Patients from 8 years old and older subjected to a variety of surgical procedures with pain of intensity at least 5/10 will be randomized into two groups: Magnetic therapy or Placebo.

The devices will be placed around the surgical wound for 2 hours. Every ten minutes, patients will rate their pain intensity on a 0-10 numerical rating scale, and morphine will be administered until pain intensity is ≤ 4/10. Pain intensity will be the primary outcome. Opioid requirements and opioid side effects will be secondary outcomes.

To detect a difference of 1 unit (from 0 to 10) between the groups with 80% power, assuming that the baseline pain intensity is 7.9 ± 2.0, we estimated the need for 70 patients per group.

We will use an intention-to-treat analysis. To analyze the effect of the treatment on pain intensity, an analysis of repeated measures using generalized estimating equations will be used. The proportion of subjects in each group who exhibit 50% or more pain relief one hour after application of the magnetic devices and the number needed to treat will also be calculated. To analyze the effect of the treatment on opioid requirements, a difference in morphine requirements between groups two hours after placement of the magnets will be estimated. To analyze the effect of the treatment on opioid side effects, a variable that summarizes the presence of any side effect two hours after the placement of the magnets will be created, and the absolute risk difference for developing any side effect will be estimated. Ninety five percent confidence intervals will be reported.

This proposal would contribute substantially to the complementary medicine field, not only because of its scientific rigor, but also because the pain model that it evaluates strengthens the validity of the results.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized or ambulatory patients 8 years old or older subjected to surgical procedures under general anesthesia, who reported at least moderate pain.

Exclusion Criteria:

* Subjects with surgeries longer than 3 hours
* Multiple surgical wounds
* Back or craniofacial surgeries, or surgeries which required cast placement, bulky dressing or the implantation of metallic devices.
* Subjects who did not understand the pain scales employed

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164
Dates: Start 2004-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity at rest

SECONDARY OUTCOMES:
Opioid requirements
Opioid side effects

CONTACTS AND LOCATIONS:
Overall Officials: M. Soledad Cepeda, MD, PhD, Principal Investigator — Javeriana University School of Medicine
Locations (1):
- San Ignacio Hospital, Bogotá, DC, Colombia

REFERENCES:
- [Result] Cepeda MS, Carr DB, Sarquis T, Miranda N, Garcia RJ, Zarate C. Static magnetic therapy does not decrease pain or opioid requirements: a randomized double-blind trial. Anesth Analg. 2007 Feb;104(2):290-4. doi: 10.1213/01.ane.0000230613.25754.08. PMID 17242082